CLINICAL TRIAL: NCT02871986
Title: Variability of Uterine and Breast Development in Response to Exogenous Oestrogen During Induction of Puberty in Individuals With Hypogonadism.
Brief Title: Pubertal Induction in Individuals With Hypogonadism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 199997
Record Dates: First submitted 2016-07-26; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-06

CONDITIONS: Primary Amenorrhoea; Hypothalamic Amenorrhoea; Hypogonadotrophic Hypogonadism; Hypopituitarism; Turner's Syndrome; Primary Ovarian Insufficiency
MeSH Terms: conditions — Hypogonadism; Hypopituitarism; Turner Syndrome; Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Individuals with hypogonadism: Individuals with hypogonadism requiring pubertal induction. Participants will receive oestrogen therapy in the form of transdermal oestrogen patch, which is standard care.
  Interventions: Drug: Routine transdermal oestrogen patch

INTERVENTIONS:
Drug: Routine transdermal oestrogen patch — Transdermal oestrogen patch will be used with an incremental dose increase at 4 months

SUMMARY:
The investigators wish to explore the variability of uterine, breast and bone outcome markers as surrogates to assess the adequacy of exogenous oestrogen replacement in individuals with hypogonadism.

DETAILED DESCRIPTION:
The investigators will invite individuals with hypogonadism who require pubertal induction to participate in the study. The participants will receive conventional routine oestrogen replacement in the form of transdermal patch. The participants will be reviewed every 2 months for a total of 8 months to document uterine, breast and bone assessment. This will be completed using a variety of tools. After 4 months, the participants will receive an incremental increase in oestrogen dose.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of hypogonadism (Turner's syndrome, hypogonadotrophic hypogonadism, primary ovarian insufficiency, hypopituitarism, hypothalamic amenorrhoea, transgender)
2. ≥ 10 years of age
3. Oestrogen naïve i.e. no prior commencement of oestrogen treatment
4. Breast Tanner stage ≤ than 2

Exclusion Criteria:

1. Previous oncology treatment
2. Primary amenorrhoea secondary to chronic medical comorbidity
3. PCOS diagnosis

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with hypogonadism requiring pubertal induction
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Uterine dimensions and volume | Assessment every 2 months for a total of 8 months
  transabdominal ultrasound

SECONDARY OUTCOMES:
Pubertal assessment - Tanner staging | Assessed every 2 months for a total of 8 months
  Conventional tanner staging
Breast Volume assessment | Assessed every 2 months for a total of 8 months
  3d Breast scanning
Height | Assessed every 2 months for a total of 8 months
  Height assessed in metres
Hormonal profile and bone turnover markers | Assessed every 2 months for a total of 8 months
  blood tests
Bone health | Assessed at baseline and at 8 months
  Routine DEXA scan
Inter and intra observer reproducibility of uterine and ovarian measurements in transabdominal ultrasound | Assessed once during the 8 month study period
  Repeat assessment by another observer
Weight | Assessed every 2 months for a total of 8 months
  Weight measured in kg
BMI | Assessed every 2 months for a total of 8 months
  BMI in kg/m^2 (weight measured in kg and height in metres)
Waist and hip circumference | Assessed every 2 months for a total of 8 months
  Measured in mm
Body fat composition | Assessed every 2 months for a total of 8 months
  Measured using standard Tanita

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Conway, FRCP, MD, Principal Investigator — UCL
Locations (1):
- University College London Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Peer Review Journals

REFERENCES:
- [Derived] Burt E, Yasmin E, Davies MC, Creighton S, Brain C, Ruff C, Learner HI, Williams L, Cameron-Pimblett A, Talaulikar V, Conway G. Variability of response to early puberty induction demonstrated by transverse uterine diameter measurement and a novel method of 3D breast imaging. Clin Endocrinol (Oxf). 2022 Jul;97(1):91-99. doi: 10.1111/cen.14740. Epub 2022 Apr 22. PMID 35436365